CLINICAL TRIAL: NCT02386865
Title: Risk Factors Predicting Prognosis and Outcome of Elderly Patients With Isolated Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Julian Joestl, MD, Medical University of Vienna
Other Study IDs: 1/2008
Record Dates: First submitted 2015-03-06; First posted 2015-03-12 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Although several prognostic models have been developed to predict outcome for patients with severe traumatic brain injury (TBI), currently no study describes the impact of respiratory failure during Emergency Department treatment on mortality in a population of elderly patients. The purpose of the present study was to evaluate factors predicting poor outcome with special emphasis on the impact of respiratory failure on mortality in elderly patients with isolated severe TBI.

All elderly patients (age ≥ 65 years) with isolated severe head injury, admitted to this Level I trauma center, during a period of 16 years (from January 1992 to December 2008) were identified from the trauma registry. Stepwise logistic regression analysis was used to identify risk factors for a poor prognosis and outcome.

The logistic regression found the following variables influencing the mortality: respiratory failure (p<0.0005; OR: 9.369), pupillary response (p<0.0212, OR: 3.393) and ISS score (p<0.0001, OR:1.179). A significant (p<0.0001) increased risk of death was also found for patients with a midline shift >15 mm.

The present study predicts a strong correlation between respiratory failure, pathological pupillary response, a higher ISS and substantial midline shift with poor outcomes in elderly patients sustaining an isolated severe TBI.

ELIGIBILITY:
The inclusion criteria for this study were:

1. patients aged 65 years and older and
2. acute severe TBI defined by an Abbreviated Injury Scale (AIS-head) score of ≥ 3 for the head region.

Exclusion criteria for this study were as followed:

1. oral intubation prior to ED-admission;
2. no details of the time of injury (e.g. chronic subdural hematomas) and
3. any concomitant injuries.
4. Patients who received oral intubation prior to ED-admission were excluded due to the high variability of indications other than respiratory failure or secondary neurological decline (e.g. intubation required for aspiration protection) that may not be necessarily related to TBI induced secondary respiratory failure.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: : All elderly patients (age ≥ 65 years) with isolated severe head injury, admitted to this Level I trauma center, during a period of 16 years (from January 1992 to December 2008) were identified from the trauma registry. Stepwise logistic regression analysis was used to identify risk factors for a poor prognosis and outcome.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Emergency Department Management | 16 years
  Interventions, Critical Care Procedures, Blood units, e.g. that were done within the first 3 hours after trauma within the emergency trauma room

SECONDARY OUTCOMES:
Glasgow Outcome Scale | 16 years

REFERENCES:
- [Derived] Ostermann RC, Joestl J, Tiefenboeck TM, Lang N, Platzer P, Hofbauer M. Risk factors predicting prognosis and outcome of elderly patients with isolated traumatic brain injury. J Orthop Surg Res. 2018 Nov 3;13(1):277. doi: 10.1186/s13018-018-0975-y. PMID 30390698